CLINICAL TRIAL: NCT03498261
Title: A Prospective Randomized Double Blind Trial to Assess the Effect of a Single Preoperative Dose of Gabapentin on Postoperative Opioid Consumption in Patients Undergoing Rhinoplasty
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Leslie Kim, Assistant Professor - Clinical, Ohio State University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2017H0466
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Adult patients scheduled to undergo rhinoplasty at the Ohio State University Wexner Medical Center
Who Masked: Participant, Investigator
Masking Description: Once the randomization group has been defined, the pharmacist will prepare both medications and will place them inside a bag for further handling. Medications will be identified following institutional standard of procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Active Comparator): The primary outcome of interest will be used to evaluate the efficacy of a single preoperative dose of gabapentin when compared to placebo on opioid consumption in patients undergoing rhinoplasty.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): The primary outcome of interest will be used to evaluate the efficacy of a single preoperative dose of gabapentin when compared to placebo on opioid consumption in patients undergoing rhinoplasty.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Gabapentin — Gabapentin has been commonly used as an adjuvant in the treatment of neuropathic pain.
  Other Names: Neurotin
  Arms: Gabapentin
Drug: Placebos — Placebo
  Arms: Placebo

SUMMARY:
Adding a single preoperative dose of gabapentin to the standard pain regimen will reduce postoperative opioid consumption within the first 72 hours in patients undergoing rhinoplasty.

DETAILED DESCRIPTION:
Study Design A prospective randomized double blind study will be conducted to assess the effect of a single preoperative dose of gabapentin on postoperative opioid consumption within the first 72 hours when compared to oral placebo in patients undergoing rhinoplasty at The Ohio State University Wexner Medical Center.

Preoperative Period After assessing patients' eligibility on the day of the surgery and written informed consent is obtained, subjects will be randomized into two groups: placebo group (group I) and gabapentin group (group II).

Pain level will be assessed and recorded at baseline using the verbal NPRS. A single dose of study medication will be administered within 2 hours before scheduled surgery time. Patients randomized to group I will receive matched oral placebo whereas patients randomized to group II will receive 900 mg of oral gabapentin. Once provided by pharmacy, the study medication will be administered by a blinded nurse in the preoperative area.

Intraoperative Period General anesthesia with desflurane and fentanyl will be provided in all patients. Other anesthetic procedures including intraoperative monitoring, muscle relaxation, endotracheal intubation, mechanical ventilation, fluid management, and the use of intravenous dexamethasone will be carried out in accordance with standard procedures. Ondansetron (4 mg) will be used as PONV prophylaxis in all patients 30 minutes before the end of the surgery. Moreover, an orogastric tube (OGT) will be used for stomach emptying at the end of the surgery and before the emergence of anesthesia.

Postoperative period Closure time will be recorded as T0. The time elapsed from PACU arrival until the first opioid dose (either oral or IV) will be recorded. Once in PACU, patients will receive IV fentanyl as pain rescue medication if required and PACU length of stay will be also recorded. After patients are considered stable based on clinician assessment and willingness to start oral intake, a treatment with oral acetaminophen 650 mg scheduled every 6 hours and oral oxycodone (5-10 mg) as needed (PRN) will be initiated for all patients.

Anesthesiologists and researchers evaluating postoperative outcomes will be blinded. The verbal NPRS will be used to assess postoperative pain level at PACU arrival, and every 30 minutes until hospital discharge. After discharge, pain levels will be recorded by patients in their diary at T6, T12, T24 (6, 12, and 24 hours after T0 respectively), and before requiring breakthrough medication (oxycodone) until postoperative day (POD) 7.

Follow-up phase Patients will be discharged home as per standard of care with oral acetaminophen 650 mg scheduled every 6 hours and a prescription for oral oxycodone 5-10 mg every 4 hours as needed (PRN). At discharge, the patient will be instructed to record his oral opioid consumption (oxycodone) and NPRS scores before each oxycodone dose until POD 7 (see attached diary).

A follow-up visit will be matched with the standard postsurgical visit at POD 7 in order to collect the diary, and count the remaining pills from the oxycodone bottle. Adverse events (AEs) including nausea and vomiting will be assessed and documented during the whole study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients males and females ≥ 18 years old
* Patients providing a written informed consent in English language
* Patients scheduled to undergo rhinoplasty under general endotracheal anesthesia

Exclusion Criteria:

1. Patients with known allergies to medications described in this study: acetaminophen, gabapentin, and opioids (morphine, fentanyl, hydromorphone, oxycodone)
2. Patients with chronic use of opioids due to any medical/surgical condition or those receiving any opioid medication within the 48 hours before surgery
3. Use of gabapentin and/or pregabalin within the last 14 days prior to surgery
4. Use of acetaminophen within the last 7 days prior to surgery
5. Hepatic disease as documented in patient past medical history
6. Medical history of autoimmune/neurodegenerative disease
7. Pregnancy or breast feeding
8. Patients with history of alcohol or substance abuse/dependency within the last 6 months
9. Patients with previous participation in this study or receiving any investigational product within the last 30 days
10. Patients under legal protection or prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Effects of Gabapentin vs Placebo in Postoperative Opioid Consumption | 72 hours
  To assess the effect of a single preoperative dose of gabapentin on postoperative opioid consumption within the first 72 hours when compared to oral placebo in patients undergoing rhinoplasty.

SECONDARY OUTCOMES:
Pain Assessment | 7 days
  To assess postoperative pain based on verbal Numeric Pain Rating Scale (NPRS), zero being no pain and ten being the worst possible pain, in the post-anesthesia care unit (PACU) and upon discharge.
IV Opioids in PACU | 7 days
  To compare intravenous opioid consumption during PACU stay
Time to rescue medication | 7 days
  To determine the time elapsed from PACU arrival until the first dose of postoperative pain rescue medication requested by the patient
Opioids within 7 days | 7 days
  To compare opioid consumption and NPRS within the first 7 days after the surgery
Length of stay (minutes) in recovery from end of surgery until discharge. | 7 days
  To assess the post-anesthesia care unit length of stay (minutes) from end of the surgery until the end of recovery phase II
Nausea | 7 days
  To compare the incidence of postoperative nausea and vomiting during PACU stay
Side Effects | 7 days
  To assess the incidence of gabapentin-related side effects
Respiratory Distress | 7 days
  To assess the incidence of respiratory distress during post-anesthesia care unit stay, defined as oxygen saturation ≤ 92%

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Kim, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishii LE, Tollefson TT, Basura GJ, Rosenfeld RM, Abramson PJ, Chaiet SR, Davis KS, Doghramji K, Farrior EH, Finestone SA, Ishman SL, Murphy RX Jr, Park JG, Setzen M, Strike DJ, Walsh SA, Warner JP, Nnacheta LC. Clinical Practice Guideline: Improving Nasal Form and Function after Rhinoplasty Executive Summary. Otolaryngol Head Neck Surg. 2017 Feb;156(2):205-219. doi: 10.1177/0194599816683156. PMID 28145848
- [Background] Demirhan A, Tekelioglu UY, Akkaya A, Bilgi M, Apuhan T, Karabekmez FE, Bayir H, Kurt AD, Kocoglu H. Effect of pregabalin and dexamethasone addition to multimodal analgesia on postoperative analgesia following rhinoplasty surgery. Aesthetic Plast Surg. 2013 Dec;37(6):1100-6. doi: 10.1007/s00266-013-0207-0. Epub 2013 Sep 21. PMID 24057811
- [Background] Sari E, Simsek G. Comparison of the Effects of Total Nasal Block and Central Facial Block on Acute Postoperative Pain, Edema, and Ecchymosis After Septorhinoplasty. Aesthetic Plast Surg. 2015 Dec;39(6):877-80. doi: 10.1007/s00266-015-0565-x. Epub 2015 Sep 22. PMID 26395094
- [Background] Wittekindt D, Wittekindt C, Schneider G, Meissner W, Guntinas-Lichius O. Postoperative pain assessment after septorhinoplasty. Eur Arch Otorhinolaryngol. 2012 Jun;269(6):1613-21. doi: 10.1007/s00405-011-1854-x. Epub 2011 Dec 1. PMID 22130915
- [Background] Argoff CE. Recent management advances in acute postoperative pain. Pain Pract. 2014 Jun;14(5):477-87. doi: 10.1111/papr.12108. Epub 2013 Aug 15. PMID 23945010
- [Background] Han B, Compton WM, Blanco C, Jones CM. Prescription Opioid Use, Misuse, and Use Disorders in U.S. Adults. Ann Intern Med. 2018 Mar 6;168(5):383-384. doi: 10.7326/L17-0700. No abstract available. PMID 29507965
- [Background] Sanders JG, Dawes PJ. Gabapentin for Perioperative Analgesia in Otorhinolaryngology-Head and Neck Surgery: Systematic Review. Otolaryngol Head Neck Surg. 2016 Dec;155(6):893-903. doi: 10.1177/0194599816659042. Epub 2016 Jul 26. PMID 27459955
- [Background] Turan A, Memis D, Karamanlioglu B, Yagiz R, Pamukcu Z, Yavuz E. The analgesic effects of gabapentin in monitored anesthesia care for ear-nose-throat surgery. Anesth Analg. 2004 Aug;99(2):375-8, table of contents. doi: 10.1213/01.ANE.0000136646.11737.7B. PMID 15271709
- [Background] Kazak Z, Meltem Mortimer N, Sekerci S. Single dose of preoperative analgesia with gabapentin (600 mg) is safe and effective in monitored anesthesia care for nasal surgery. Eur Arch Otorhinolaryngol. 2010 May;267(5):731-6. doi: 10.1007/s00405-009-1175-5. Epub 2009 Dec 10. PMID 20012076
- [Background] Helander EM, Billeaud CB, Kline RJ, Emelife PI, Harmon CM, Prabhakar A, Urman RD, Kaye AD. Multimodal Approaches to Analgesia in Enhanced Recovery After Surgery Pathways. Int Anesthesiol Clin. 2017 Fall;55(4):51-69. doi: 10.1097/AIA.0000000000000165. No abstract available. PMID 28901981
- [Background] Mathiesen O, Dahl B, Thomsen BA, Kitter B, Sonne N, Dahl JB, Kehlet H. A comprehensive multimodal pain treatment reduces opioid consumption after multilevel spine surgery. Eur Spine J. 2013 Sep;22(9):2089-96. doi: 10.1007/s00586-013-2826-1. Epub 2013 May 17. PMID 23681498